CLINICAL TRIAL: NCT07159347
Title: Assessment of Stressors in Children With Depressive Symptoms for the Development of an App to Strengthen Emotional Competences Using Serious Games and Gamification.
Brief Title: Assessment of Daily Stressors in Children With Depressive Symptoms for the Development of a Gamified Emotion Regulation App
Acronym: SG4ChildD
Status: Recruiting | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Technical University Darmstadt (WG Serious Games) (Unknown); Ascora GmbH (Unknown); smart medication eHealth Solutions GmbH (Unknown); Pedagogical Academy Elisabethenstift gGmbH (Unknown); University Medical Center Rostock (Other); Johannes Gutenberg-University Mainz (Developmental Psychology) (Unknown); Federal Ministry of Research, Technology and Space (Unknown)
Responsible Party: Principal Investigator, Ellen Greimel, Principal investigator, Ludwig-Maximilians - University of Munich
Other Study IDs: 25-0508
Record Dates: First submitted 2025-08-27; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Depressive Disorder; Depression in Children; Depressive Symptoms
Keywords: depression; daily hassles; qualitative interviews; focus groups; serious gaming; gamification; participatory needs assessment; emotion regulation skills
MeSH Terms: conditions — Depressive Disorder; Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- children aged 8-12 years with increased depressive symptoms: This cohort includes children aged 8-12 years who report increased depressive symptoms based on a questionnaire. Participation involves a semi-structured interview on daily hassles and self-report questionnaires on stress perception and emotion regulation. No intervention is provided.
- parents of children aged 8-12 years with increased depressive symptoms: This cohort includes parents of children with increased depressive symptoms aged 8-12. Parents take part in a focus group to discuss their child's exposure to daily hassles, coping strategies and ways their child can be supported. They also complete self-report questionnaires. No intervention is provided.

SUMMARY:
Digital interventions, such as serious games, are becoming increasingly important in the context of prevention and treatment approaches of mental disorders. A project (SG4ChildD) funded by the Federal Ministry of Research, Technology and Space (BMFTR) aims to develop a gamified app to promote emotion regulation in children aged 8 to 12 with increased depressive symptoms or a manifest diagnosis of depression. The app intends to train emotion regulation skills through playful and everyday-relevant scenarios. To ensure that the app meets the needs of the target group, a participatory needs assessment will be conducted that involves both children and their parents. Based on interviews with children and focus groups with parents and complemented by questionnaires, it will be assessed which everyday stressors children experience, how they cope with them, and what kind of support they and their parents find helpful.

DETAILED DESCRIPTION:
Depressive disorders are among the most common psychiatric disorders in youth. Early depression can have serious effects on psychosocial development and long-term life outcomes. Despite the high demand for early intervention, substantial barriers to care persist, including long waiting times for therapy and administrative obstacles. As a result, low-threshold, location-independent interventions play an increasingly important role in improving access to care. In recent years, digital interventions such as serious games have gained increasing recognition in this context. These purposefully designed digital games go beyond mere entertainment by delivering targeted health-promoting, therapeutic, or psychoeducational content.

An important therapeutic focus in childhood depression is the improvement of emotion regulation - an ability strongly linked to mental health and resilience. The overarching goal of the present BMFTR-funded research project (SG4ChildD) is the development of a gamified app aimed at strengthening emotion regulation skills in children aged 8 to 12 with increased depressive symptoms or depressive disorders, serving as an add-on to professional treatment. In the current subproject, a participatory needs assessment with the app's target group (children with increased depressive symptoms/depressive disorders) and their parents will be conducted prior to the development of the app.The subproject aims to gain a deeper understanding of (1) everyday stressors experienced by children with depressive symptoms, (2) the subjective perception and emotional impact of these stressors, (3) the coping strategies children apply, and (4) the parental perspective on children's emotional challenges and supportive needs.

For this purpose, a primarily qualitative approach is chosen. Following an initial screening questionnaire to assess eligibility, participating children will take part in a semi-structured interview focusing on their subjective experience of emotional stress in everyday life (daily hassles). The interview will e.g. explore situations that trigger sadness or frustration and examine how children attempt to manage these feelings. This will be supplemented by standardized questionnaires on daily hassles, stress exposure and emotion regulation. In parallel, focus groups will be conducted with parents to explore their observations regarding children's exposure to daily hassles, coping strategies and what kind of support they and their children might need. Additionally, parents will complete questionnaires assessing their own regulatory parenting skills (i.e., the degree to which parents assist their children in the use of different regulation strategies) and parental report of the child´s depressive symptoms.

The insights gained through this needs assessment will directly inform the development of the app, and particularly the selection of game-based scenarios that reflect children's real-world challenges. By involving children and parents at an early stage of development, the project aims to maximize usability, acceptance, and clinical relevance of the digital intervention.

Participants will be recruited based on predefined inclusion criteria (e.g., elevated depressive symptoms in children). Recruitment will primarily take place via the Department of Child and Adolescent Psychiatry, Psychosomatics, and Psychotherapy at the LMU University Hospital Munich. Additional recruitment may be supported by collaborating child and adolescent psychiatric clinics in the Munich area and by licensed outpatient therapists.

ELIGIBILITY:
Inclusion Criteria (Children):

* increased depressive symptoms indicated by either (1) self report assessed with Beck Depression Inventory for Youth 2 (Beck et al., 2019; T-score > 60) , or (2) parental report assessed with DISYPS-III - external rating scale for depressive disorders (FBB-DES; Döpfner et al., 2017; applying gender- and age-normed Stanine scores ≥ 7).

Exclusion Criteria (Children):

* Insufficient German language skills
* Acute suicidality
* Schizophrenic disorder
* Severe developmental disorder
* Mental and behavioral disorders due to psychotropic substances

Inclusion Criteria (Parents):

Parent of a child meeting the above inclusion criteria

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: In total, 15-20 participants will be included in the study, including both children aged 8-12 with increased depressive symptoms and parents of children with increased depressive symptoms. Parents will be included in the study (focus group), even if their child is not taking part in the study and vice versa. The sample size is based on the concept of data saturation, which refers to the point at which no new information emerges from additional data.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Qualitative data from semi-structured child interviews and parental focus groups | Start of appointment, after questionnaire on depressive symptoms
  Data will be collected through semi-structured individual interviews with children and focus group discussions with parents. The aim is to explore children's exposure to daily hassles, the subjective perception and emotional impact of these hassles, coping strategies, and support needs.

SECONDARY OUTCOMES:
Daily Hassles (Child-Report) | During the Appointment, after semi-structured interview
  Assessed with the German translation of the Daily life stressors Scale (Kearney et al., 1993)
Perceived Stress (Child-Report) | During the Appointment, after semi-structured interview
  Assessed with the German translation of the Perceived stress scale - children (White, 2014)
Emotion regulation strategies (Child-Report) | During the Appointment, after semi-structured interview
  Assessed with the Process-Oriented Emotion Regulation Questionnaire for Children and Adolescents (Rüth & Lohaus, 2023)
Regulatory parenting skills (parental report) | During the Appointment, after focus group
  German translation of the Parental Assistance with Child Emotion Regulation (Cohodes et al., 2022)

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Schulte-Körne, Prof. Dr., Principal Investigator — Department of Child and Adolescent Psychiatry, Psychosomatics and Psychotherapy, LMU University Hospital; Ellen Greimel, Prof. Dr., Principal Investigator — Department of Child and Adolescent Psychiatry, Psychosomatics and Psychotherapy, LMU University Hospital
Locations (1):
- Department of Child and Adolescent Psychiatry, Psychosomatics and Psychotherapy, LMU University Hospital, München, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No
The data collected in this study include sensitive details about participants, such as various sociodemographic and clinical characteristics. Publicly sharing the raw dataset could risk revealing individual identities, thereby violating ethical standards related to participant confidentiality. As a result, the data will not be publicly released. However, detailed descriptions of the methodology, materials used, and sample characteristics will be provided within the article and supplementary materials. Aggregated data and additional supporting materials may be shared upon request (contact: Lisa.Feldmann@med.uni-muenchen.de).